CLINICAL TRIAL: NCT05078606
Title: Pre-anesthetic Ultrasonographic Assessment of Neck Vessels as Predictors of Spinal Anesthesia Induced Hypotension in Elderly: a Prospective Observational Study.
Brief Title: Ultrasonographic Assessment of Neck Vessels as Predictors of Spinal Anesthesia Induced Hypotension in Elderly
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassant M. Abdelhamid, Associate professor, Cairo University
Other Study IDs: MD-152-2020
Record Dates: First submitted 2021-10-04; First posted 2021-10-14 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Post-spinal Hypotension
MeSH Terms: interventions — Carotid Intima-Media Thickness; Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: IJV Ultrasonography — Patient will be in supine position, The linear probe with frequency of 7- 12 M hz; depth of 3 cm. maximum IJV diameter (IJV-D) and area (IJV-A) will be recorded. M-mode will be used to obtain the distance between the 2 walls of the vein during inspiration and expiration.
  Then, the patient will be positioned 10° Trendelenburg and similar ultrasonographic measurements will be again performed
Device: Carotid Intima Media Thickness — US Probe is slided superiorly (toward the head) or inferiorly (toward the feet) until the bifurcation of the common carotid artery (CCA) appears on the left side of the screen. This is the ideal location for imaging and CIMT measurements.
  IMT is assessed in longitudinal view from the arterial far wall, along a 10mm length. CIMT will appear as two parallel lines (leading edges of two anatomical boundaries) from it: lumen- intima and media- adventitia interfaces perpendicular to ultrasound beams.
Procedure: Spinal anesthesia — Spinal anesthesia will be performed in the sitting position at level of L3-4 or L4- 5 interspaces with a 25-gauge spinal needle. Local infiltration of skin and subcutaneous tissue with 2% lignocaine will be applied. After confirming cerebrospinal fluid flow, 10 mg of 0.5% hyperbaric bupivacaine plus 25 mcg fentanyl will be injected. The degree of sensory block (cold test by alcohol gauze) will be assessed in the study with a goal of T8 dermatomal level block.

SUMMARY:
Spinal anesthesia induces sympathetic blockade and venodilation, thus reducing venous return and the cardiac output. Therefore, assessment of intravascular volume deficit before anesthesia might predict a critical decrease in blood pressure after anesthesia.

Recently, ultrasonographic evaluation of the internal jugular vein (IJV) has been used to reflect intravascular volume status and fluid and as a predictor of hypotension after induction of general anesthesia.

Carotid intima-media thickness (CIMT) has been used to predict atherosclerosis-related events, such as stroke, myocardial infarction, peripheral artery disease, and hypotension after induction of anesthesia with a cut-off value of 0.65 mm of CIMT as a threshold level.

DETAILED DESCRIPTION:
This study aims to evaluate the ability of preoperative Ultrasonographic assessment of the internal jugular vein (IJV) and Carotid intima-media thickness (CIMT) to predict spinal anesthesia induced hypotension (SAIH).

Participants will be elderly patients (above 60 years), ASA I-II-III, scheduled for elective surgeries under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>60 years)
* ASA I-II-III
* Patients scheduled for elective surgeries under spinal anesthesia.

Exclusion Criteria:

* Operations which will last for less than 15 minutes.
* Deep vein thrombosis in the upper extremities.
* History of radiotherapy or neck surgery.
* Previous sonographic data show tricuspid or mitral regurgitation or a very distended right atrium and ventricle.
* Patients with history of valvular or carotid artery surgery, arrhythmia, heart failure.
* Being unable to lie in a supine position for the necessary measurements.
* Technical limitations to imaging of the IJV and carotid artery.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be elderly patients (above 60 years), ASA I-II-III, scheduled for elective surgeries under spinal anesthesia.
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Accuracy of IJV collapsibility index as predictor of Spinal anesthesia induced hypotension. | 10 minutes
  (Area under receiver operating characteristic curves)

SECONDARY OUTCOMES:
Accuracy of rate of change in IJV area with change in posture as a predictor of Spinal anesthesia induced hypotension. | 10 minutes
  (Area under receiver operating characteristic curves)
Incidence of Spinal anesthesia induced hypotension | 20 minutes
  Change in mean arterial blood pressure 25% less than the preoperative baseline level.
Carotid intima media thickness. | 10 minutes
  IMT is measured as the distance between lumen-intima and media-adventitia interfaces
Norepinephrine consumption | 20 minutes
  the total dose of norepiniphrine and number of boluses

CONTACTS AND LOCATIONS:
Overall Officials: Bassant abdelhamid, Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Singh Y, Anand RK, Gupta S, Chowdhury SR, Maitra S, Baidya DK, Singh AK. Role of IVC collapsibility index to predict post spinal hypotension in pregnant women undergoing caesarean section. An observational trial. Saudi J Anaesth. 2019 Oct-Dec;13(4):312-317. doi: 10.4103/sja.SJA_27_19. PMID 31572075
- [Background] Pre-operative ultrasonographic evaluation of inferior vena cava collapsibility index and caval aorta index as new predictors for hypotension after induction of spinal anaesthesia: A prospective observational study: erratum. Eur J Anaesthesiol. 2019 Nov;36(11):888. doi: 10.1097/EJA.0000000000001094. No abstract available. PMID 31580292